CLINICAL TRIAL: NCT04356573
Title: (KIWI) Speeding up a Slow Protein for Muscle Mass With Hay Kiwifruit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 206814
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Metabolism; Protein

STUDY DESIGN:
Intervention Model Description: Subjects crossed over between ingesting 2 different types of kiwifruit for 2 weeks prior to each stable isotope metabolic study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Biological samples were coded and code list password protected until all data was analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gold Kiwifruit First, then Green Hayward Kiwifruit (Placebo Comparator): Subjects first ate 2 gold kiwifruit with midday meal for 2 weeks before crossing over to the green Hayward kiwifruit intervention
  Interventions: Dietary Supplement: Green Hayward Kiwifruit first, then Gold Kiwifruit; Dietary Supplement: Gold Kiwifruit First, then Green Hayward Kiwifruit
- Green Hayward Kiwifruit first, then Gold Kiwifruit (Active Comparator): Subjects first ate 2 green Hayward kiwifruit with midday meal for 2 weeks before crossing over to the gold kiwifruit intervention
  Interventions: Dietary Supplement: Green Hayward Kiwifruit first, then Gold Kiwifruit; Dietary Supplement: Gold Kiwifruit First, then Green Hayward Kiwifruit

INTERVENTIONS:
Dietary Supplement: Green Hayward Kiwifruit first, then Gold Kiwifruit — Subjects ate 2 peeled green kiwifruit with their midday meal for 2 weeks prior to testing.
Dietary Supplement: Gold Kiwifruit First, then Green Hayward Kiwifruit — Subjects ate 2 peeled gold kiwifruit with their midday meal for 2 weeks prior to testing.

SUMMARY:
The specific hypothesis is that the consumption of 2 Hayward green kiwifruit (containing actinidin protease) prior to 100g of ground beef will increase the rate of protein digestion from the beef in the elderly, leading to an increased uptake of the essential amino acids. Furthermore, this increased essential amino acid availability will produce a greater postprandial net anabolic protein response, as well as increased fractional synthetic rates of muscle proteins.

DETAILED DESCRIPTION:
The specific hypothesis is that the consumption of 2 Hayward green kiwifruit (containing actinidin protease) prior to 100g of ground beef will increase the rate of protein digestion from the beef in the elderly, leading to an increased uptake of the essential amino acids. Furthermore, this increased essential amino acid availability will produce a greater postprandial net anabolic protein response, as well as increased fractional synthetic rates of muscle proteins.

To test this hypothesis, the investigators will use a double-blinded crossover design involving two intervention arms; in both arms 100g of ground beef (cooked weight) will be consumed following either 2 Hayward green kiwifruit (containing actinidin protease) or 2 Hort16A Gold kiwifruit (devoid of actinidin protease) by elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* men and women ages 60-85 inclusive.

Exclusion Criteria:

* Inability to chew meats or difficulty swallowing solid foods
* History of diabetes
* History of malignancy in the 6 months prior to enrolment
* History of gastrointestinal reduction or bypass surgery (Lapband, etc)
* History of a chronic inflammatory condition or disease (Lupus, HIV'AIDS, etc)
* History of chronic kidney disease or currently requiring dialysis.
* Allergy to beef or kiwifruit
* Subjects who do not or will not eat animal proteins
* Subjects who cannot refrain from consuming protein or amino acid supplements during their participation in this study
* Subjects who report regular resistance exercise (more than once per week)
* Hemoglobin less than 9.5mg/dL at the screening visit
* Platelets less than <150,000 at the screening visit
* Subjects who are not willing or able to suspend aspirin for several days prior to their muscle biopsies.
* Subjects who have been prescribed a blood-thinning medication (Coumadin, lovenox, heparin, Plavix, etc).
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arny A Ferrando, Ph.D., Principal Investigator — UAMS professor
Locations (1):
- UAMS Center on Aging, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Church DD, Starck C, Schutzler SE, Azhar G, Kim IY, Ferrando AA, Moughan PJ, Wolfe RR. The impact of Hayward green kiwifruit on dietary protein digestion and protein metabolism. Eur J Nutr. 2021 Mar;60(2):1141-1148. doi: 10.1007/s00394-020-02363-5. Epub 2020 Sep 24. PMID 32970234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol enrollment was 13 participants, each was to complete 2 conditions in crossover fashion (i.e., either green kiwi followed by yellow kiwi, or yellow kiwi followed by green kiwi). One subject dropped out, which left 6 subjects in each group.
Groups:
- Gold Kiwifruit First, Then Green Hayward Kiwifruit: Subjects were first asked to eat 2 gold kiwifruit with midday meal for 2 weeks prior to testing.
  Later, subjects were asked to eat 2 green Hayward kiwifruit with midday meal for 2 weeks prior to a second set of testing.
- Green Hayward Kiwifruit First, Then Gold Kiwifruit: Subjects were first asked to eat 2 green Hayward kiwifruit with midday meal for 2 weeks prior to testing.
  Later, subjects were asked to eat 2 gold kiwifruit with midday meal for 2 weeks prior to a second set of testing.
Period: Overall Study
Arm/Group | Gold Kiwifruit First, Then Green Hayward Kiwifruit | Green Hayward Kiwifruit First, Then Gold Kiwifruit
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — Didn't Qualify | 1 | 0

BASELINE CHARACTERISTICS:
Population: 12 participants completed both crossover conditions. 1 individual failed screening.
Groups:
- Gold Kiwifruit First, Then Green Hayward Kiwifruit: Subjects were first asked to eat 2 gold kiwifruit with midday meal for 14 days prior to testing. Then a washout for 14 days. Then, subjects were asked to eat 2 green Hayward kiwifruit with midday meal for 2 weeks prior to a second set of testing.
- Green Hayward Kiwifruit First, Then Gold Kiwifruit: Subjects were first asked to eat 2 green Hayward kiwifruit with midday meal for 2 weeks prior to testing. Then a washout for 14 days. Then, subjects were asked to eat 2 gold kiwifruit with midday meal for 2 weeks prior to a second set of testing.
- Total: Total of all reporting groups
Arm/Group | Gold Kiwifruit First, Then Green Hayward Kiwifruit | Green Hayward Kiwifruit First, Then Gold Kiwifruit | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (6.2) | 72.1 (6.2) | 72.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Net Balance Measured by Gas Chromatography-Mass Spectrometry (GC-MS)
Description: Blood samples were analyzed to quantify the appearance of the stable isotopes: 2H2-tyrosine, 2H4-tyrosine, and 2H5-phenylalanine in tracer to tracee ratio or mole percent excess. Changes in these markers over time enable the calculation of whole body protein metabolism. Calculations are done as follows:
  Total plasma rate of appearance = infusion rate/enrichment Fractional rate of appearance of tyrosine from phenylalanine= 2H4-tyrosine/2H5-phenylalanine Phenylalanine hydroxylation = fractional rate of appearance of tyrosine from phenylalanine x rate of appearance of tyrosine Protein Synthesis = [(rate of appearance of phenylalanine -Phe hydroxylation) x 25] Protein Breakdown = [(rate of appearance of phenylalanine - phenylalanine infusion rate) x 25 - phenylalanine intake] Net Balance = Protein Synthesis - Protein Breakdown
Time Frame: 300 minutes
Measure: Mean (Standard Deviation); unit: g protein per 300 mins
Groups:
- Gold Kiwifruit: Subjects ate 2 gold kiwifruit with midday meal for 2 weeks.
  fresh kiwifruit: Subjects ate 2 peeled kiwifruit with their midday meal for 2 weeks prior to testing.
- Green Hayward Kiwifruit: Subjects ate 2 green Hayward kiwifruit with midday meal for 2 weeks.
  fresh kiwifruit: Subjects ate 2 peeled kiwifruit with their midday meal for 2 weeks prior to testing.
Arm/Group | Gold Kiwifruit | Green Hayward Kiwifruit
Number analyzed (Participants) | 12 | 12
g protein per 300 mins | 14.58 (4.31) | 14.55 (3.24)

2. Secondary Outcome: Change in Skeletal Muscle Protein Metabolism Measured by Gas Chromatography-Mass Spectrometry (GC-MS)
Description: Muscle samples were analyzed to quantify the appearance of the stable isotope 2H5-phenylalanine in trace to tracee ratio or mole percent excess. The change in 2H5-phenylalanine in subsequent muscle biopsy allow for the calculation of muscle protein synthesis. The calculation is done as follows: [(2H5-phenylalanine enrichment in second biopsy - 2H5-phenylalanine enrichment in second biopsy)/ (2H5-phenylalanine plasma enrichment × time)] × 60 × 100.
Time Frame: 9.5 hours
Measure: Mean (Standard Deviation); unit: % per hour
Arm/Group | Gold Kiwifruit | Green Hayward Kiwifruit
Number analyzed (Participants) | 12 | 12
% per hour | 0.0043 (0.0244) | 0.0081 (0.0393)
Statistical Analysis 1: Comparison: Gold Kiwifruit vs Green Hayward Kiwifruit; Test type: Superiority; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: While subjects were enrolled in the study; up to two months.
Groups:
- Gold Kiwifruit: Subjects ate 2 gold kiwifruit with midday meal for 2 weeks.
  Half of the subjects ate the gold kiwifruit first, half of the subjects ate the gold kiwifruit second; however all subjects ate 2 gold kiwifruit with midday meal for 2 weeks at some point in this study.
- Green Hayward Kiwifruit: Subjects ate 2 green Hayward kiwifruit with midday meal for 2 weeks.
  Half of the subjects ate the green Hayward kiwifruit first, half of the subjects ate the green Hayward kiwifruits second; however all subjects ate 2 green Hayward kiwifruit with midday meal for 2 weeks at some point in this study.
Arm/Group | Gold Kiwifruit | Green Hayward Kiwifruit
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gold Kiwifruit (N=12) | Green Hayward Kiwifruit (N=12)
Viral Bronchitis (Infections and infestations) | 1 (1) | 0 (0) — Event unrelated to study treatments/arms. Subject told staff she was diagnosed with viral bronchitis on Oct. 24th. Treated with abx on 11/9/18. Nearly resolved as of 11/20/18.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04356573/Prot_SAP_001.pdf